CLINICAL TRIAL: NCT01757990
Title: A Comparative Clinical Evaluation of the Effect of Stevia Rebaudiana Extracts and Sucrose on Dental Plaque pH (Stephan Curve Trend) Using a Microtouch Electrode in Healthy Volunteers. A Phase II Study.
Brief Title: The Effect of Stevia Rebaudiana Extracts on Different Variables Related to Caries: an in Vitro and in Vivo Evaluation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Guglielmo Campus, Associate Professor of Community Dentistry, Università degli Studi di Sassari
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SS_2012_10
Record Dates: First submitted 2012-12-22; First posted 2012-12-31 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Dental Caries
Keywords: dental caries; Stevioside; Rebaudioside; plaque pH; Streptococcus mutans
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stevioside extract (Experimental): After measuring baseline plaque pH, the subjects rinsed for 1 minute with the solution containing Stevioside extract. Plaque pH was then measured at 5, 10, 15, 30, 45 and 60 min after the mouth rinse.
  Interventions: Dietary Supplement: Effect of Stevioside and Rebaudioside on plaque pH
- Rebauside extract (Experimental): After measuring baseline plaque pH, the subjects rinsed for 1 minute with the solution containing Rebaudioside extract. Plaque pH was then measured at 5, 10, 15, 30, 45 and 60 min after the mouth rinse.
  Interventions: Dietary Supplement: Effect of Stevioside and Rebaudioside on plaque pH
- Saccarosio (Sham Comparator): After measuring baseline plaque pH, the subjects rinsed for 1 minute with the sucrose solution. Plaque pH was then measured at 5, 10, 15, 30, 45 and 60 min after the mouth rinse.
  Interventions: Dietary Supplement: Effect of Stevioside and Rebaudioside on plaque pH

INTERVENTIONS:
Dietary Supplement: Effect of Stevioside and Rebaudioside on plaque pH — After measuring baseline plaque pH, the subjects rinsed for 1 minute with the sucrose solution. Plaque pH was then measured at 5, 10, 15, 30, 45 and 60 min after the mouth rinse.

SUMMARY:
The aim of the present investigation was to evaluate the effect of stevioside and rebaudioside on several variables related to caries development. Two approaches were performed: an in vitro evaluation of the growth of a culture of mutans streptococci and in vivo randomized study on the effect of a single rinse containing stevioside and rebaudioside on plaque-pH.

ELIGIBILITY:
Inclusion Criteria:

good general health, normal salivary secretion rate, normal buffer capacity

Exclusion Criteria:

systemic diseases, salivary secretion reduction, reduced buffer capacity

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Plaque-pH modification | 5, 10, 15, 30, 45, 60 minutes
  Plaque pH was measured at baseline and 5, 10, 15, 30, 45 and 60 minutes after each mouth rinse

CONTACTS AND LOCATIONS:
Overall Officials: Laura Strohmenger, MD, Study Chair — WHO Collaborating Centre for Community Dentistry and Oral Epidemiology University of Milan